CLINICAL TRIAL: NCT01246739
Title: Adrenalectomy Versus Follow-up in Patients With Mild Hypercortisolism: a Prospective Randomized Controlled Trial
Brief Title: Adrenalectomy Versus Follow-up in Patients With Subclinical Cushings Syndrome
Acronym: AUSC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010/297
Record Dates: First submitted 2010-11-18; First posted 2010-11-23 (Estimated); Last update posted 2024-04-10 (Actual); Status verified 2024-03

CONDITIONS: Adrenal Tumour With Mild Hypercortisolism
Keywords: mild hypercortisolism; adrenal tumour; surgical procedures, elective; indication
MeSH Terms: conditions — Adrenal Gland Neoplasms | interventions — Adrenalectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Follow-up (No Intervention): Patients who are diagnosed with biochemically mild hypercortisolism (so-called subclinical Cushing´s syndrome), who are followed only.
- Surgery (Experimental): Patients diagnosed with adrenal tumour and with biochemically mild hypercortisolism (so-called subclinical Cushing´s syndrome), operated with adrenalectomy
  Interventions: Procedure: Adrenalectomy

INTERVENTIONS:
Procedure: Adrenalectomy — Adrenalectomy (open or laparoscopic)
  Arms: Surgery

SUMMARY:
Incidental findings of adrenal tumours,"incidentalomas", occur in 1-5 % in the general population and 10-25 % of these patients will exhibit biochemical mild hypercortisolism. Although the patients do not have clinical signs of classical Cushing's syndrome, they have an increased risk for hypertension, dyslipidemia, diabetes mellitus, osteoporosis and obesity.

The hypothesis of the study is, that surgery of the adrenal adenoma responsible for the increased secretion of cortisol, will in part cure or ameliorate the metabolic syndrome.

DETAILED DESCRIPTION:
Adrenal incidentalomas, adrenal tumours detected without symptoms and signs of hormonal hypersecretion or malignancy, are common. Depending on modality (MRI, CT. Ultrasonography) adrenal tumours occur in approximately 1-5% of the population. In about 10% of patients, the tumours are bilateral. At autopsy studies adrenal tumours occur in 1% of patients under the age of 30, but in approximately 7% of patients older than 70 years. Investigation of the adrenal tumours focus on to exclude malignancy (which is uncommon), and an increased secretion of hormones (adrenaline, aldosterone, cortisol), so-called functional tumours. However, most often adrenal incidentalomas are non-functional. The most common functional disorder is increased secretion of cortisol, and then usually without clinical stigmata, known as subclinical Cushing's syndrome (or mild hypercortisolism). Clinical stigmata, Cushing's syndrome, is empirically associated with elevated levels of urinary cortisol.

Subclinical Cushing's syndrome occurs in 10-25% of patients with adrenal incidentalomas. The incidence has been estimated at 0.8 / 1,000 inhabitants, making it a common disease.

Diagnosis is based to detect an autonomous release of cortisol from the adrenal gland (a disorder of the so-called hypothalamic-pituitary-adrenal axis).

Fundamental to the diagnosis is that the secretion of cortisol is not inhibited <50 nmol / L at 8.00, after an overnight test with 1 mg of oral dexamethasone.

In addition, at least one of the following criteria for disturbance of the hypothalamic-pituitary-adrenal axis is suggested to be present:

* attenuated or abolished circadian rhythm of cortisol
* ACTH in the low normal range or supressed
* DHEAS low or supressed (age dependent)

Numerous studies have shown that high blood pressure, diabetes, impaired glucose tolerance, and unfavourable lipid profile, is common in patients with subclinical Cushing's syndrome, and basically do not differ from patients with overt Cushing's syndrome. At follow-up of patients with adrenal incidentalomas, some patients exhibit intermittent mild hypersecretion of cortisol, others develop overt Cushing's syndrome (unusual) and still some patients with initially normal hypothalamic-pituitary-adrenal axis, develop a subclinical Cushing's syndrome.

The aim of this study is to investigate if adrenalectomy for subclinical Cushing's syndrome (mild hypercortisolism without clinical signs), result in an improvement in cardiovascular risk factors, cardiac function, and arteriosclerosis compared to follow-up

ELIGIBILITY:
Inclusion Criteria:

* Adrenal tumour with biochemical mild hypercortisolism defined as pathological dexamethasone suppression test (cortisol > 50 nmol/L at 8.00 am after 1 mg dexamethasone at 10 pm, plus one of the following criteria

  * Low or suppressed adrenocorticotropic hormone (ACTH)
  * Low or suppressed dehydroepiandrosterone (DHEA)
  * No or pathological circadian rhythm of cortisol

Exclusion Criteria:

* Increased levels of 24 hours urinary excretion of cortisol
* Pregnancy or lactation
* Inability to understand information or to comply with scheduled follow-up
* Mild hypercortisolism with bilateral adrenal tumours, without a gradient (lateralization on venous sampling)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-06; Primary Completion 2024-02 (Actual); Study Completion 2024-02 (Actual)

PRIMARY OUTCOMES:
Improvement of blood pressure as assessed by 24 hours blood pressure measurement | At two years after intervention
  Blood pressure assessed by 24 hours measurement is considered to be improved if at least one of the following outcomes has occurred, and is sustained, during 2 years of follow-up:
  1. Normalization of hypertension without medical treatment
  2. Unchanged or decreased blood pressure in patients with hypertension if the number or dose of the patient's antihypertensive drug (s) has been reduced
  3. Unchanged normal blood pressure in patients who were normotensive at the time of randomization.

SECONDARY OUTCOMES:
Normalization of diabetes mellitus | At two years after intervention
  Normalization of diabetes mellitus according to the criteria of the World Health Organization and assessed by oral glucose tolerance test
Decreased body mass index (BMI) to < 30 | At two years post intervention
  Standard assessment of BMI
Bone density | At two years post intervention
  Bone density assessed with dual energy x-ray absorptiometry (DEXA) at the lumbar spine and hip
Blood lipids | At two years post intervention
  Triglyceride and cholesterol changes of whole serum and of the lipoprotein classes; low-density-lipoprotein (LDL), very-low-density-lipoprotein (VLDL) and high-density-lipoprotein (HDL)
Cardiac function | At two years post intervention
  Cardiac function assessed by echocardiography; left ventricular ejection fraction (EF), left ventricular end-diastolic diameter (LVDD), left ventricular mass index (LVMI), ratio between mitral peak velocity flow of the early filling wave and the atrial wave (E/A ratio)
Cognitive function | At two years after intervention
  Mini Mental State Examination (MMSE) for cognitive function
Quality of Life assessed by SF 36 | At two years after intervention
  Quality of Life assessed by the generic instrument short form 36 (SF-36).
Atherosclerosis | At two years after intervention
  Carotid ultrasound/duplex scans with evaluation of intimal thickness and plaques.
  Blood pressure measurement for ankle index
Adrenal cortical insufficiency | At two years after intervention
  Rate of patients with postoperative adrenal cortical insufficiency in patients operated due to subclinical Cushings syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Anders OJ Bergenfelz, MD, PhD, Principal Investigator — Department of Surgery, Skåne University Hospital, Lund, Sweden
Locations (4):
- Århus University Hospital, Aarhus, Denmark
- Haukeland University Hospital, Bergen, Norway
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Skåne University Hospital-Lund, Department of Surgery, Lund

REFERENCES:
- [Derived] Ueland GA, Ragnarsson O, Heie A, Kjellbom A, Lindgren O, Muth A, Palazzo F, Poulsen PL, Rolighed L, Thordarson HB, Wernig F, Bergenfelz A. Randomized trial studying metabolic outcomes and quality of life after adrenalectomy versus conservative management for mild autonomous cortisol secretion. Endocr Connect. 2025 Jul 19;14(7):e250361. doi: 10.1530/EC-25-0361. Print 2025 Jul 1. PMID 40600855